CLINICAL TRIAL: NCT02672566
Title: Low-molecular-weight Heparin in Constituted Vascular Intrauterine Growth Restriction. Randomized Multicenter Trial
Brief Title: Low-molecular-weight Heparin in Constituted Vascular Intrauterine Growth Restriction
Acronym: GROWTH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1508175; 2016-000424-25 (EudraCT Number)
Record Dates: First submitted 2016-01-28; First posted 2016-02-03 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2019-04

CONDITIONS: Fetal Growth Retardation
Keywords: Fetal Growth Retardation; enoxaparin
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Enoxaparin; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group : enoxaparin (Experimental): Experimental group will take enoxaparin (4000 Ui / Day) and will benefit from the usual care.
  Interventions: Drug: Enoxaparin; Other: Usual care
- Control group (Active Comparator): The control group will only benefit from the usual care.
  Interventions: Other: Usual care

INTERVENTIONS:
Drug: Enoxaparin — Enoxaparin will be delivered to the patients every day at the dose of 4 000 Ui.
  Other Names: Treatment
  Arms: Experimental group : enoxaparin
Other: Usual care — Patients will all benefit from the usual care
  Other Names: Classic support

SUMMARY:
Intrauterine growth restriction (IUGR) is correlated to an abnormal placenta development, with an alteration of the maternal-fetal circulation, coagulation troubles, and apparition of placental infarcts. IUGR represents the third cause of perinatal mortality in France, and is associated to an important morbidity. For birth-weights < 10th percentile of the gestational age, the neonatal death risk is doubled, compared to abnormal weights. In 35% of cases, IUGR is of vascular origin and is included in the broader framework of placental vascular pathology (PVP).

Up to now, studies have focused on the primary or secondary prevention of PVP. Few studies have evaluated the treatment of constituted vascular IUGR. Currently, the management of vascular IUGR is mainly based on active surveillance, or termination of pregnancy. Pathological findings suggest that placental pro-thrombotic phenomena play a role in the constitution of vascular IUGR. Since aspirin is not effective in reducing this type of event, a randomized, open-label study conducted in China compared 14-day treatment with low-molecular-weight heparin (LMWH) versus Dan-Shen (a product not used in France) after diagnosis of IUGR. This trial, including 73 patients, showed a significant improvement in average growth kinetics in the LMWH group. The mean birth weight was 2877 g in the heparin group and 2492 g in the Dan-Shen group (p <0.0001). However, no data were provided concerning the number of newborns with a birth weight <10th percentile, i.e. the risk of morbidity and mortality, or complications occurring. Due to the lack of reliable data, LMWH are not included in the currently recommended therapeutic strategy for vascular IUGR.

The studies in IUGR reported to date mainly focused on primary or secondary prevention in women at risk of PVP, assessing the value of aspirin, which showed only a modest effect. No effective therapeutic strategy is available to treat patients with constituted vascular IUGR, a situation where LMWH should be more effective than antiplatelets given the vascular context.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years being at a gestational age ≥ 22 and <34 weeks of gestation with vascular fetal growth retardation defined according CNGOF
* Ultrasound Estimated fetal weight below the 10th percentile
* Clinical and ultrasound findings suggesting pathologically impaired growth or diminished foetal well-being
* Clinical and ultrasound findings suggesting placental insufficiency
* Precise dating of pregnancy with an ultrasound between 11 + 0 and 13 + 6 weeks of gestation
* Written informed consent

Exclusion Criteria:

* multiple pregnancy or identified cause of IUGR (intra-uterine growth retardation)
* Patient with an immediate indication of fetal extraction
* Women with a history of venous thromboembolism or already treated with anti-coagulant
* Women with a contraindication to enoxaparin treatment at prophylactic doses
* Patient refusing to participate or unable to consent
* Patient with less than 80,000 platelets / mm 3 with the initial assessment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Number of new born with a weight inferior at the 10th percentile | Week 36
  With the AUDIPOG formula, the number of new born with a weight inferior at the 10th percentile will be calculated.

SECONDARY OUTCOMES:
Change in doppler parameters of uterine arterie | baseline from delivery
  Doppler parameters is a composite outcome : pulsatility index and presence of notch
Change in doppler parameters of ombilical arterie | baseline from delivery
  Doppler parameters is a composite outcome : resistance index, presence of a zero diastole or reverse flow
Change in doppler fetal weight | baseline from delivery
  doppler fetal weight (grams)
birth weight | delivery
  birth weight (grams)
Number of new born with a weight inferior at the 3rd percentile | delivery
  With the AUDIPOG formula, the number of new born with a weight inferior at the 3rd percentile will be calculated.
Number of fetal extraction | before 36 weeks of gestation
  fetal extraction
number of major neonatal parameters | 1 month after delivery
  Major neonatal parameters is at least one or more : Perinatal death, Ischemic encephalopathy Major intra- or periventricular bleeding (grade 3 or 4), Periventricular leukomalacia, Necrotizing enterocolitis, Bronchopulmonary dysplasia or Sepsis
number of minor neonatal parameters | 1 month after delivery
  Minor neonatal parameters is a composite outcome : Caesarean section for fetal distress, Cord arterial pH < 7.1, Apgar score <7 at 5 minutes
Number of Major bleeding events (MB) and clinically relevant non-major bleeding events (CRNMB) | from randomisation to 1 month postpartum
  The definitions of major bleeding events and clinically major bleeding events are adapted from the ISTH definition for which were added a specific Obstetrics and Gynaecology definition Bleeding events (MB) is a composite outcome.
Number of thrombocytopenia | From randomisation to 36 weeks
  thrombocytopenia is a composite outcome : Thrombopenia defined by platelet count < 100 G/L Significant thrombocytopenia with HIT suspicion defined as follows:≥ 40% decline of the platelet count (compared with baseline value) occurring during the first 8 weeks following the start of HBPM Or platelet count < 80 Giga/l to terme

CONTACTS AND LOCATIONS:
Overall Officials: Tiphaine Raia-Barjat, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (8):
- France (8):
  - Chru Brest, Brest
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Chu Grenoble, Grenoble
  - Ch Lyon Sud Pierre Benite, Lyon
  - HFME - Lyon Est, Lyon
  - Hopital Croix Rousse Lyon, Lyon
  - Ch Roanne, Roanne
  - Chu Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No